CLINICAL TRIAL: NCT06506175
Title: A Phase I Clinical Trial to Evaluate the Effects of Different Dosing Conditions, Timing and Food on the Pharmacokinetics of HRS9531 Tablets in Healthy Subjects
Brief Title: Investigation of Optimal Dosage Regimen for HRS9531 Tablets in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS9531-T-102
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Overweight or Obese, Type 2 Diabetes
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Comparisons between arms with different dosing conditions, timing and food for oral HRS9531 tablets
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Treatment group A：Different fasting time、dosing conditions and timing (Experimental)
  Interventions: Drug: HRS9531 tablets
- Treatment group B：Different fasting time、dosing conditions and timing (Experimental)
  Interventions: Drug: HRS9531 tablets
- Treatment group C：Different fasting time、dosing conditions and timing (Experimental)
  Interventions: Drug: HRS9531 tablets
- Treatment group D：Different fasting time、dosing conditions and timing (Experimental)
  Interventions: Drug: HRS9531 tablets
- Treatment group E：Different fasting time、dosing conditions and timing (Experimental)
  Interventions: Drug: HRS9531 tablets
- Treatment group F：Different fasting time、dosing conditions and timing (Experimental)
  Interventions: Drug: HRS9531 tablets
- Treatment group G：Fed conditions (Experimental)
  Interventions: Drug: HRS9531 tablets
- Treatment group H：Fasting conditions (Experimental)
  Interventions: Drug: HRS9531 tablets

INTERVENTIONS:
Drug: HRS9531 tablets — HRS9531 tablets

SUMMARY:
The study is being conducted to evaluate the effects of different dosage regimen on the pharmacokinetics of HRS9531 tablets in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the trial procedures, be able and willing to provide a written informed consent.
2. Male subject aged 18-55 years (both inclusive) at the time of signing informed consent.
3. Body weight ≥50.0 kg, body mass index (BMI) of 24.0-35.0 kg/m^2 (both inclusive) at screening.
4. Weight change does not exceed 5 kg within 3 months before screening.
5. Good general health as judged by the investigator, based on medical history, physical examination, vital signs, clinical laboratory and electrocardiogram (ECG).

Exclusion Criteria:

1. Known or suspected hypersensitivity to trial product(s) or related products.
2. With previous major organ diseases, including but not limited to neuropsychiatric, cardiovascular, digestive, respiratory, urinary, endocrine, blood, immune and other diseases, are judged by researchers to be unsuitable for the study.
3. Abnormal and clinically significant blood pressure at screening.
4. History of significant gastrointestinal diseases or related symptoms (e.g., nausea, vomiting, heartburn, or diarrhea), conditions affecting gastric emptying (e.g., pyloric stenosis), or previous gastrointestinal surgery (excluding polypectomy and appendectomy), or acute diarrhea or constipation within 7 days before randomization.
5. Blood donation within 1 month prior to screening, or blood donation ≥400 mL or blood loss ≥400 mL within 3 months prior to screening.
6. Presence of any clinically significant results in examination at screening visit.
7. Hepatitis B surface antigen (HBsAg), HIV antibody detection, treponema pallidum specific antibody detection, hepatitis C virus antibody (HCVAb) positive.
8. Presence of - clinically significant ECG results.
9. Known or suspected history of drug abuse or drug abuse, or urine drug screening test during the screening periodThose who are positive.
10. Addiction to tobacco and alcohol.
11. Individuals with special dietary habits deemed unsuitable for participation by the investigator, or those unable to adhere to the dietary requirements of the trial during the study period.
12. In the opinion of the investigator, there are any other conditions that interfere with the evaluation of the results of the trial or are not suitable for participation of this study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-08-05 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
AUCtau | 0-24hrs after the 10th dosing
  Area under the HRS9531 tablets concentration curve from time 0-24 hours after the 10th dosing

SECONDARY OUTCOMES:
Tmax | First dose at day 1 and post-dose at day 10
  Time to maximum plasma concentration
Cmax | First dose at day 1 and post-dose at day 10
  The maximum plasma concentration
t1/2 | First dose at day 1 and post-dose at day 10
  Terminal half-life
Incidence and severity of adverse events | Screening period up to Day 45
Anti-HRS9531 antibody | Before First dose at day 1 to Day 45

CONTACTS AND LOCATIONS:
Locations (1):
- The affiliated hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided